CLINICAL TRIAL: NCT05149248
Title: Prevention and Control of Neoplasms Associated With HPV in High-risk Groups in Mexico City: The Condesa Study
Acronym: CONDESA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); National Council of Science and Technology, Mexico (Other)
Responsible Party: Principal Investigator, Eduardo Cesar Lazcano Ponce, Deputy Director, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SECITI/094/2017
Record Dates: First submitted 2021-09-18; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Cancer of Cervix
Keywords: NEOPLASMS; HPV; PREVENTION; CONTROL; HIGH RISK
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18; Vaccines, Synthetic; Control Groups

STUDY DESIGN:
Intervention Model Description: This study is a mixed methods study combining public health interventions offering primary and secondary prevention of HPV to populations highly vulnerable to these health problems with evaluation of the interventions in a 12-month follow-up. In addition, the study includes qualitative interviews that will undergo systematic analysis on the perceptions, meanings, and individual experiences of the intervention, within the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1: MSM (Other): Arm 1: HPV vaccination in an alternative schedule for MSM of 1 dose (M0). Arm 2: HPV vaccination in an alternative schedule for MSM of 2 doses over a 6-month period (M0,6) Arm 3: a control group will be screened for high-risk HPV and vaccinated at 12 months
  Interventions: Biological: Gardasil® [Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant vaccine]; Biological: Two dose; Other: Control group
- Group 2: TRANSGENDER WOMEN (Other): Arm 1: Transgender women
  Interventions: Biological: 2 dose vaccination over 6 month
- GROUP 3: WOMEN AND MEN LIVING ON THE STREET (Other): Arm 1: Women and men living on the street
  Interventions: Biological: 2 dose vaccination over 6 month
- GROUP 4: WOMEN AND MEN WHO HAVE SUFFERED RAPE (Other): Women and men who have suffered rape
  Interventions: Biological: 2 dose vaccination over 6 month
- GROUP 5: WOMEN WHO ARE SEX WORKERS (Other): Female sex workers
  Interventions: Biological: 2 dose vaccination over 6 month

INTERVENTIONS:
Biological: Gardasil® [Quadrivalent Human Papillomavirus (Types 6,11,16,18) Recombinant vaccine] — HPV vaccination in an alternative schedule for MSM of 1 dose (M0).
  Arms: Group 1: MSM
Biological: Two dose — HPV vaccination in an alternative schedule for MSM of 2 doses over a 6-month period (M0,6)
  Arms: Group 1: MSM
Other: Control group — HPV vaccination at 12 months
  Arms: Group 1: MSM
Biological: 2 dose vaccination over 6 month — 2-dose HPV vaccination regimen over a 6-month period (M0,6)
  Arms: GROUP 3: WOMEN AND MEN LIVING ON THE STREET; GROUP 4: WOMEN AND MEN WHO HAVE SUFFERED RAPE; GROUP 5: WOMEN WHO ARE SEX WORKERS; Group 2: TRANSGENDER WOMEN

SUMMARY:
Objective: To evaluate the effectiveness of a combined strategy of human papillomavirus virus (HPV) vaccination and high-risk HPV screening to reduce the occurrence of neoplasms in the anogenital region and oral cavity among men who have sex with men, people with HIV, homeless people, transgender women, female sex workers and rape victims.

Methods: This mixed methods study evaluates the effectiveness of a combined vaccination-screening strategy to reduce HPV prevalence/incidence and occurrence of cervical intraepithelial neoplasms grade 2+ and/or anal intraepithelial neoplasms grade 2+, using Kaplan-Meier. The time-to-event method will evaluate time from positive results for specific anogenital HPV to incidence of anogenital lesions containing that HPV type.

Conclusions: This study will generate scientific evidence on effectiveness of a combined vaccination-screening strategy to reduce the burden of HPV-associated neoplasms within vulnerable populations in Mexico.

DETAILED DESCRIPTION:
Men who have sex with men (MSM), people with HIV, homeless people (many of whom participate in survival sex), female sex workers, transgender women and rape victims are at high risk for human papillomavirus (HPV) infection and consequently developing cancers associated with chronic HPV infection including cervical, vaginal , vulvar , and anal cancers in women, cancer of the penis , anal cancer, in men, and cancer of the oropharynx , tongue, and tonsils in both men and women, In part, this is related to increased life expectancy among people with HIV (given greater anti-retroviral treatment coverage).

Some countries have implemented HPV vaccination policies that include men. This is based on promotion of protection against an increased risk of HPV infection, universal increase in coverage and a gender equity perspective . Since population-level introduction of HPV vaccines, there has been a dramatic impact in areas with over 60% vaccination coverage. Decreases of approximately 90% have been reported for HPV-6/11/16/18 infections, over 90% for new cases of genital warts, 45% for low-grade cytological abnormalities, and 85% for anogenital high-grade histological lesions .

The HPV FASTER concept combines HPV vaccination with HPV screening. It is based on the HPV vaccine's high efficacy and the high sensitivity of high-risk HPV testing for primary detection of anogenital cancer precursor lesions (as documented by our research group in more than 200,000 Mexican women). This strategy is effective because HPV vaccination among women and men over a wide age range offers protection to those not currently infected and protects against subsequent re-infections16. Thus, a combined HPV vaccination and screening strategy will potentially: 1) mitigate the demand for timely screening tests by expanding screening intervals; 2) improve the cost-benefit balance of secondary prevention programs; and 3) provide greater protection and quality of life to more people by reducing the burden of diseases attributable to HPV. This intervention can save many lives over the next 30 years and be more cost-effective than traditional approaches.

Recently, the US vaccination advisory group recommended HPV vaccination among sexually abused children, recognizing their increased risk of HPV infection , . The US Centers for Disease Control recommends administering the HPV vaccine to subjects with immunosuppressive conditions, HIV infection, and men who have sex with men . HPV vaccination in HIV-positive people is safe and reduces the incidence of HPV-associated cancers, including anal cancer, which is increasing in these populations , . Moreover, some research has shown that vaccination against HPV in populations with HIV is cost-effective.

HPV serotypes 16 and 18, found in the HPV bivalent and tetravalent vaccines, have an estimated relative contribution to invasive cervical cancer of at least 70% in Latin America. These vaccines are highly effective, provide high levels of immunogenicity , have acceptable security profiles and have been incorporated into public vaccination policies with 3-dose schedules over a 6-month period based on pharmaceutical industry recommendations.

Alternative schedules of population vaccinations have been implemented in spite of the conflict of interest with the pharmaceutical industry. The first of these schedules was conducted in Quebec, Canada where the extended 0-6-60 month schedule was promoted for girls under 16 years . Later, in Mexico, a similar vaccination program recommended by a group of experts coordinated by the National Institute of Public Health was initiated. Mexico was a pioneer in adopting a 2-dose alternative vaccination schedule in April 2014. Currently, there is evidence that alternative schedules are not inferior to the traditional schedule in terms of immunogenicity . In 2012 , Switzerland adopted a 2-dose vaccination schedule against HPV in girls under 15 years old under assuming age was the main mediator of the protection induced by the vaccine and not the number of doses. This assumption would explain why the vaccine was the main inducer of IgG responses, plasma cells, and memory B cell formation and why 2 doses administered with a 6-month interval provided similar protection during the initial years of vaccination.

In April 2014, the Council officially pronounced the adoption of a vaccination schedule against HPV with only 2 doses with a periodicity of 0 and 6 months. The justification for this resolution, in which Mexico was a pioneer and was subsequently officially recommended by the WHO as a vaccination policy at a global level, was that the immunological responses of girls aged 9 to 11 years after two doses of HPV vaccine were similar to or greater than those obtained after three doses in women aged 16 to 26 years.

The benefits of this decision are logistical and economic; increasing coverage and providing greater flexibility in the application of the second dose. Moreover, the savings generated from not administering a third dose are considerable. Alternative schedules with two doses and schedules with a third dose at 60 months in girls 9-11 years of age can offer a) improvements in the immune response in the medium- and long-term, because there is evidence that a new exposure to HPV increases the expression of antibodies logarithmically, and b) advantages in its administration, since it is easier to organize these schedules within the framework of schools and consequently provides a better opportunity for equity in obtaining greater coverage and adherence to complete schedules in the captive population before leaving compulsory schooling. However, although the recommendation is plausible from an immunological perspective, there is no evidence from clinical trials of efficacy to support this determination for ethical reasons.

Currently, a paradigm shift is perceived toward the application of a single dose of vaccine against HPV. Research groups at a global level are evaluating the hypothesis that men and women who receive one versus two doses do not have a higher prevalence of HPV and that consequently the effect of the intervention is equivalent.

In this regard, demonstration studies are being conducted in population universes to evaluate the effect of a single dose of HPV vaccine. The strategy is to evaluate the effect of administering 1 versus 2 doses in a specific community using a randomized intervention allocation strategy. In the 2-dose intervention group, the most biologically and logistically efficient approach is to administer the second intervention between 6 and 12 months after the first intervention. The outcome to be evaluated in men who have sex with men is the presence of HPV DNA in the anal canal, which is obtained and determined in the basal measurement during the administration of the first dose. This type of intervention is feasible in Mexico due to its invaluable tradition of innovation in public policies for the prevention and control of anogenital cancer and its implementation of large demonstration studies. Currently, it can be affirmed that with the current evidence, vaccination of all groups at risk of anogenital cancer with a single dose will be the preamble to the attenuation of the impact of persistent HPV infections and their consequent lesions .

Methods Hypotheses

* The application of a combined HPV vaccination scheme and screening through the identification of high-risk HPV subtypes will reduce the prevalence of HPV infection in the oral and anogenital cavities in the different study groups, at 12 months post-vaccination. Consequently, the occurrence of grade 2 or higher anal intraepithelial neoplasia (AIN 2+) lesions in men and high-grade or higher cervical intraepithelial neoplasia (CIN 2+) lesions in women will decrease.
* Alternative vaccination schedules of one versus two doses of prophylactic vaccines against HPV are equivalent in terms of effectiveness.
* Urine and self-collected vaginal, anal canal, and oral cavity samples constitute an alternative epidemiological surveillance approach for monitoring the impact of a combined strategy HPV vaccination and screening for high-risk HPV subtypes in vulnerable populations.

Objectives Primary objective

• To evaluate the effectiveness of a combined strategy of HPV vaccination and screening for high-risk HPV subtypes to reduce the occurrence of HPV in the anogenital region and oral cavity in five highly vulnerable groups in Mexico City, Mexico: men who have sex with men, female sex workers, transgender women, subjects living in street situations, and people who have suffered rape.

Secondary objectives

* To evaluate the effectiveness of alternative HPV vaccination schedules.
* To evaluate the usefulness of the collection of self-collected vaginal, anal, and urine samples as alternatives for monitoring the impact of a combined strategy of HPV vaccination and screening based on the detection of high-risk HPV subtypes.
* To assess the barriers to and facilitators of the introduction of a combined HPV vaccination and primary screening strategy with tests for high-risk HPV subtypes in the study groups.

Study population and procedures The sample sizes for the five cohorts are: 6,000 MSM, 500 transgender women, 400 homeless men and women, 400 sexual assault victims, 2500 female sex workers. This study is a mixed methods study combining public health interventions offering primary and secondary prevention of HPV to populations highly vulnerable to these health problems with evaluation of the interventions in a 12-month follow-up. In addition the study includes qualitative interviews that will undergo systematic analysis on the perceptions, meanings, and individual experiences of the intervention, within the study groups.

A central element of the present project is a parallel study of five sentinel cohorts of the adult population ≥ 14 years and ≤ 45 years of age that is operationally coordinated by the Condesa and Iztapalapa Specialized Clinics, which belong to the health services of Mexico City and the Program of Care for rape victims. This program is coordinated by the Specialized Clinics in collaboration with the Mexico City Attorney General of Justice.especially the Victims Care Center, which is a program of the Center for Therapy in Support of Victims of Sex Crimes. The investigators attempt to include at least 80% of the population of each interest group in the epidemiological component of the project. Study subjects will be recruited (2018-2019) during their routine care within any program or service the participant attend within the Condesa and Iztapalapa Specialized Clinics; in addition, posters will be placed within the clinics inviting potential study subjects to participate and civil society organizations which collaborate with the clinics will be visited regularly to invite persons involved in their activities to participate in the study.

For the qualitative intervention component, individuals from the five vulnerable groups will be selected for voluntary participation in qualitative semi-structured interviews. This sub-sample will be purposely selected to include the maximum variation of characteristics, and 12 to 16 semi-structured individual interviews will be conducted for each study group. These interviews will explore perceptions of HPV, experiences as users of preventive care for HPV and related cancers, acceptability of and meanings related to HPV vaccination and barriers to and facilitators of primary prevention (vaccination) and secondary prevention (screening and treatment) of HPV.

The study protocol and instruments were approved by the Research, Ethics and Biosecurity Committees of the National Institute of Public Health. All study participants will provide signed informed consent before participating in any study procedure or completing any study instruments (and consent forms will be signed by two witnesses).

Sample collection and vaccination At the beginning of the study, all MSM who agree to participate in the study will receive the HPV vaccination in an alternative schedule for MSM of 1 versus 2 doses over a 6-month period. In addition, a control group will be screened for high-risk HPV and vaccinated at 12 months. For transgender women, women and men living on the street, and women and men who have suffered rape, a 2-dose regimen of the tetravalent HPV vaccine will be administered over a 6-month period. The additional combined strategy corresponds to screening for high-risk HPV subtypes to identify intraepithelial lesions in the transformation zone of the anal and/or cervical canals.

Additionally, samples will be self-collected from the anal canal, oral cavity, and vaginal canal. These samples will be collected both at the baseline measurement and at 12 months after vaccination to assess changes in the prevalence and incidence of new HPV infections in the different study groups. All HPV-positive anal and cervical samples will be evaluated using liquid-based cytology; analysis will be done at the National Institute of Public Health.

On a single occasion, additional samples will be collected from a proportional sample of the different study groups (70% of MSM and 90% of women, not including transgender women) for the identification of other STIs, including Neisseria gonorrhea, syphilis, HIV, herpes simplex virus type 2, hepatitis B virus, and hepatitis C virus. Positive cases will be referred to the corresponding medical care within their respective affiliated clinics.

The HPV detection test has been installed at the National Institute of Public Health with the Cobas 4800 HPV platform. This test is a qualitative test that detects 14 high-risk genotypes using specific probes. It detects genotypes 16 and 18 individually and a pool of other types (31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66, and 68) cataloged as high risk.

Cytological evaluation will be conducted for all HPV-positive samples from both the anal canal and cervix. A urine sample will be obtained, centrifuged, and prepared for DNA extraction. The sample will be stored at -20°C prior to processing for HPV detection. The techniques for these purposes are under evaluation. Blood samples (10-ml) will be collected from the study participants by vacuum venipuncture. The collected samples will be centrifuged to separate the sera into 2-ml aliquots, which will be stored in cryo-vials at -20°C prior to processing. Antibody responses to viral and bacterial etiological agents will be conducted as follows:

* Hepatitis B and hepatitis C. Automated enzyme-linked immunosorbent assay. The analytical procedure will be conducted according to the corresponding manufacturer's laboratory instructions , .
* Syphilis. The Venereal Disease Research Laboratory (VDRL) screening test and the Serodia Treponema pallidum (TP) confirmatory test by particle agglutination. The analytical procedures will be performed in accordance with the laboratory instructions of the corresponding manufacturers .
* Herpes simplex virus type 2. Microplate immuno-enzymatic assay for the detection of type-specific viral antibodies. Confirmation of positive samples by Western blotting assay. The analytical procedures will be performed in accordance with the laboratory instructions of the corresponding manufacturers In cervical samples, an automated chemo-luminescent assay for bacterial DNA detection will be performed using polymerase chain reaction (PCR). The analytical procedure will be conducted according to the corresponding manufacturer's laboratory instructions .

Data analysis To estimate the effectiveness of the strategy of combining HPV vaccination with HPV screening, the differences in the prevalence of HPV and the cumulative incidence of HPV infection and/or development of CIN 2+ and/or AIN 2+ will be estimated during the first 12 months of follow-up using the Kaplan-Meier method. The time-to-event method will be applied to evaluate the time from the specific type of HPV genital positivity to the incidence of anogenital lesions harboring the same HPV subtype within the lesion. The analytical unit for this study is HPV 16/18 type-specific infection and generic high-risk strain infection.

The transcripts of individual interviews will be analyzed with through coding transcribed material, which implies the classification of pieces of the interviews into a priori and emerging categories to systematize the information and search for patterns, similarities, and differences.

ELIGIBILITY:
Inclusion Criteria:

* Between 14 and 45 years of age
* Men who identify themselves as having sex with other men
* Transgender women
* Women or men living on the street/homeless
* Women or men who have suffered rape
* People with or without HIV infection

Exclusion Criteria:

* Under 14 years or over 45 years of age
* History of any serious adverse reaction prior to any component of the influenza vaccine, such as life-threating, hospitalization, partial or total disability, or incurable damage
* Chronic HIV infection in stages A3, B3 and C3, and/or CD4 cell count less than 200 cells per cubic millimeter
* Presence in the HIV-positive participant of an active opportunistic infection such as: Toxoplasma Gondii encephalitis, Cryptococcosis, Tuberculous meningitis, Pulmonary tuberculosis, Community acquired pneumonia, Pneumocystis jiroveci, Isosporidiasis, Cryptosporidiasis, Salmonellosis, Candida esophagitis and esophagitis, Esophagitis Vascular neoplasia
* Pregnancy confirmed by laboratory test
* Previous vaccination against HPV
* Previous treatment of intraanal lesions

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6000 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
HPV DNA in anal, vaginal, and oral cavity. | 18 months to achieve 12-month follow-up in group 1 MSM
  Change in prevalence of any and specific HPV DNA in anal, vaginal and oral cavity from baseline and at 12 months after vaccination.

SECONDARY OUTCOMES:
Prevalence of any and specific HPV DNA in anal, vaginal and oral cavity at 12 months after vaccination between groups | 18 months to achieve 12-month follow-up in group 1 MSM and competition of all the interviews
  Change in prevalence of any and specific HPV DNA in anal, vaginal and oral cavity at 12 months after vaccination between groups
Invalid results in each self-collected sample type: vaginal, anal and urine | 18 months to achieve 12-month follow-up in group 1 MSM
  Number of invalid results in each self-collected sample type: vaginal, anal and urine
Barriers to and facilitators of the introduction of a combined HPV vaccination and primary screening strategy with tests for high-risk HPV subtypes in the study groups. | Up to 18 months
  For the qualitative intervention component, individuals from the five vulnerable groups will be selected for voluntary participation in qualitative semi-structured interviews. This sub-sample will be purposely selected to include the maximum variation of characteristics, and 12 to 16 semi-structured individual interviews will be conducted for each study group. These interviews will explore perceptions of HPV, experiences as users of preventive care for HPV and related cancers, acceptability of and meanings related to HPV vaccination and barriers to and facilitators of primary prevention (vaccination) and secondary prevention (screening and treatment) of HPV. The transcripts of individual interviews will be analyzed with through coding transcribed material, which implies the classification of pieces of the interviews into a priori and emerging categories to systematize the information and search for patterns, similarities, and differences.

OTHER OUTCOMES:
Secondary prevention of the STIs included in this project will be achieved among individuals belonging to vulnerable groups who are the target population of this intervention. | 18 months to achieve 12-month follow-up in group 1 MSM
  Number of positive cases to Neisseria gonorrhea, syphilis, HIV, herpes simplex virus type 2, hepatitis B virus, and hepatitis C virus in a subsample of 70% of MSM and 90%of women, not including transgender women). Positive cases will be referred to the corresponding medical care within their respective affiliated clinics

CONTACTS AND LOCATIONS:
Overall Officials: EDUARDO C LAZCANO PONCE, PHD, Principal Investigator — Instituto Nacional de Salud Publica, Mexico
Locations (1):
- Instituto Nacional de Salud Publica, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263